CLINICAL TRIAL: NCT00683098
Title: Long-term Results After Endoscopic Total Extraperitoneal Repair of Recurrent Inguinal Hernia
Status: Completed | Type: Observational
Sponsor: St. Claraspital AG (Other)
Responsible Party: Principal Investigator, Urs Pfefferkorn, Surgical Registrar, St. Claraspital AG
Other Study IDs: TEP Clara
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Hernia
Keywords: recurrent hernia; endoscopic total extraperitoneal repair; inguinal pain; questionnaire
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: patients, who had a endoscopic total extraperitoneal repair of recurrent inguinal hernia between 1995 and 2008

SUMMARY:
Evaluation of long-term results for chronic pain and impairment of daily activities after endoscopic total extraperitoneal repair of recurrent inguinal hernia with inguinal pain questionnaire (IPQ).

DETAILED DESCRIPTION:
Evaluation of long-term results for chronic pain and impairment of daily activities after endoscopic total extraperitoneal repair of recurrent inguinal hernia with inguinal pain questionnaire (IPQ).

All patients, who had a endoscopic preperitoneal mesh repair of a recurrent inguinal hernia between 1995 and 2008 were prospectively recorded and will be sent the IPQ via mail.

ELIGIBILITY:
Inclusion Criteria:

* patients, who had endoscopic total extraperitoneal repair of recurrent inguinal hernia at our institution between 1995 and 2008

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients, who had endoscopic total extraperitoneal repair of recurrent inguinal hernia at our institution between 1995 and 2008
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2008-06; Primary Completion 2008-08 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Pain according to Inguinal Pain Questionnaire Activity according to Inguinal Pain Questionnaire | up to 10 years

SECONDARY OUTCOMES:
Recurrence, Reoperation | up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Urs Pfefferkorn, MD, Principal Investigator — Department of Surgery
Locations (1):
- St. Claraspital, Basel, Switzerland

REFERENCES:
- [Background] Staarink M, van Veen RN, Hop WC, Weidema WF. A 10-year follow-up study on endoscopic total extraperitoneal repair of primary and recurrent inguinal hernia. Surg Endosc. 2008 Aug;22(8):1803-6. doi: 10.1007/s00464-008-9917-9. Epub 2008 Apr 29. PMID 18443875
- [Background] Hallen M, Bergenfelz A, Westerdahl J. Laparoscopic extraperitoneal inguinal hernia repair versus open mesh repair: long-term follow-up of a randomized controlled trial. Surgery. 2008 Mar;143(3):313-7. doi: 10.1016/j.surg.2007.09.028. Epub 2008 Jan 14. PMID 18291251
- [Background] Franneby U, Gunnarsson U, Andersson M, Heuman R, Nordin P, Nyren O, Sandblom G. Validation of an Inguinal Pain Questionnaire for assessment of chronic pain after groin hernia repair. Br J Surg. 2008 Apr;95(4):488-93. doi: 10.1002/bjs.6014. PMID 18161900